CLINICAL TRIAL: NCT03899519
Title: The Correlations of the Findings Obtained From Airway Ultrasonography With Cormack Lehane Classification in Patients With Obstructive Sleep Apnoea - A Cross Sectional Study
Brief Title: Airway Ultrasonography Measurements With Cormack Lehane Classification in Patients With OSA
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Senior Consultant Anaesthetist and Lecturer, Universiti Sains Malaysia
Other Study IDs: USM/JEPeM/18010094
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea; Difficult Intubation
Keywords: OSA; ultrasound; airway; difficult intubation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Airway assessment using ultrasonography can provide an additional information in identifying difficult intubation in OSA patients. The main purpose of this study is to find the correlation of the ultrasound parameters and the Cormack Lehane Score (CL Score) as well as to identify the cut-off point of the ultrasound parameters that would differentiate between the easy and difficult intubation.

DETAILED DESCRIPTION:
Research design

1. This is a cross sectional study. Involving face-to-face interview, USG airway assessment and Cormack Lehane score assessment. The patient will be identified from locations listed below:

   * Anaesthesia clinic
   * In the ward, during review by anaesthesia team for elective operation in the following day
   * In the ward, when cases are notified for operations as emergency case
2. Once consent obtained from the patient, information regarding surgery and date of surgery will be recorded in the patient's data collection sheet. Patient's STOPBANG score and AHI score will also be recorded.
3. The airway ultrasonography will be performed by the principal investigator using a standardized ultrasound machine (NextGen LOGIC e Ultrasound with 12L-RS wide band linear array 5-13 MHz frequency probe) under supervision by a radiologist. The procedure will be performed at the recovery bay in the operation theatre. The following measurements will be done and recorded for future statistical analysis.

   * Depth of preepiglottic space (PE)
   * Distances between epiglottis and midpoint between 2 vocal cords (E-VC)
4. Cormack Lehane score will be obtained during induction of General Anaesthesia and Intubation in OT on the specified OT date. Conventional direct laryngoscope will be used for CL score determination. Medical Officer of more than 2 years' experiences in anaesthesiology will be requested to intubate the patient to minimize bias. CL scores are as described below

CL 1: Most of glottis Visible CL 2: Half of the glottis seen CL 3: Only epiglottis visible CL4: No laryngeal structure visible

Study area: Hospital Sultanah Nurzahirah, Kuala Terengganu Study population: Adult patient age between 18 to 65, diagnosed or suspected OSA, planned for operation under General Anaesthesia

Sample size estimation

1. st Objective :

   * To determine the correlation between airway ultrasonography measurements and CL score.
   * Using R package pwr

     * For PE

       * r: 0.595 (based on Gupta D, 2012), significant level 0.05, power: 0.8
       * Number of sample: 19
     * For E-VC

       * r: -0.966 (based on Gupta D,2012), significant level 0.05, power: 0.8)
       * Number of sample: 4
     * For ratio PE/E-VC

       * r: 0.495 (based on Gupta D, 2012), significant level 0.05, power: 0.8)
       * Number of sample: 28
2. nd and 3rdobjective

   * 2nd objective: To determine the best cut off point of airway ultrasonography measurement in predicting the difficulty in intubation using CL (difficult vs less difficult)
   * 3rd objective: To determine the accuracy of cut-off point in determining difficult intubation. (AUC) )
   * Receiver Operating characteristics (ROC) curve power calculation using R

     * Significance level: 0.05
     * Power of study: 0.8
     * Kappa: 4
     * AUC: 0.7

Based on previous study, the incidence of difficult intubation in OSA patient is 19.3%. Hence kappa: 4. Using pROC package in R, based on the above values and data, the investigators need at least 24 cases of difficult intubation and 41 cases of non-difficult intubation (to detect AUC of 0.7 from 0.5 null hypothesis). So, total patients required is at least 65

Sampling method and subject recruitment As mentioned above, this is a cross sectional study. Involving face-to-face interview, USG airway assessment and Cormack Lehane score assessment. After the samples identified at the specific locations mentioned and they will be approached for consent. Once agreed, the patient will be recruited for the study.

Data analysis

Statistical Analysis Plan For objective 1

• Intended statistical analysis: Spearman correlation

For objective 2 and 3

* Using ROC curve
* outcome: difficulty status (0 or 1)
* test variable: PE, E-VC and ratio PE/E-VC

AUC in the ROC curve will be calculated accordingly based on the study results

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65
2. Diagnose / screened OSA
3. Planned for operation under General Anaesthesia
4. American Society Of Anaesthesia (ASA) physical status class I-III

Exclusion Criteria:

1. Unstable haemodynamic status
2. Patient refusal to participate
3. Altered mental status, cognitive function or mental disorder
4. Distorted head and neck anatomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patient age between 18 to 65, diagnosed or suspected OSA, planned for operation under General Anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation between airway ultrasonography measurements and CL score | may 2017-may 2018
  ultrasound measurements
Cut off point of airway ultrasonography measurement in predicting the difficulty in intubation using CL | may 2017-may 2018
  ultrasound measurements
Accuracy of each cut off point in objective 2 | may 2017-may 2018
  cut off point to differentiate between easy and difficult intubation

CONTACTS AND LOCATIONS:
Overall Officials: Rhendra Hardy Mohamed Zaini, Principal Investigator — University Sains Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta D, Srirajakalidindi A, Ittiara B, Apple L, Toshniwal G, Haber H. Ultrasonographic modification of Cormack Lehane classification for pre-anesthetic airway assessment. Middle East J Anaesthesiol. 2012 Oct;21(6):835-42. PMID 23634565
- [Result] Rana S, Verma V, Bhandari S, Sharma S, Koundal V, Chaudhary SK. Point-of-care ultrasound in the airway assessment: A correlation of ultrasonography-guided parameters to the Cormack-Lehane Classification. Saudi J Anaesth. 2018 Apr-Jun;12(2):292-296. doi: 10.4103/sja.SJA_540_17. PMID 29628843
- [Result] Soltani Mohammadi S, Saliminia A, Nejatifard N, Azma R. Usefulness of Ultrasound View of Larynx in Pre-Anesthetic Airway Assessment: A Comparison With Cormack-Lehane Classification During Direct Laryngoscopy. Anesth Pain Med. 2016 Aug 15;6(6):e39566. doi: 10.5812/aapm.39566. eCollection 2016 Dec. PMID 28975073